CLINICAL TRIAL: NCT00980239
Title: A Multi-arm Phase I Trial of Hepatic Arterial Infusion of Irinotecan With 1) Systemic Bevacizumab 2) Systemic Bevacizumab and Oxaliplatin 3) Systemic Bevacizumab and Cetuximab in Patients With Advanced Cancers Metastatic to the Liver
Brief Title: HAI Irinotecan + IV Bevacizumab, Bevacizumab & Oxaliplatin or Bevacizumab & Cetuximab in Advanced Cancers Metastatic to Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0410; NCI-2012-01272 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-09-17; First posted 2009-09-21 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Liver Cancer; Advanced Cancer
Keywords: Solid Tumors; Liver; hepatic arterial infusion; HAI; Bevacizumab; Avastin; Cetuximab; Erbitux; Irinotecan; Camptosar; Oxaliplatin; Eloxatin
MeSH Terms: conditions — Liver Neoplasms | interventions — Irinotecan; Bevacizumab; Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Group 1 = Irinotecan + Bevacizumab
  Interventions: Drug: Irinotecan; Drug: Bevacizumab
- Group 2 (Experimental): Group 2 = Irinotecan, Bevacizumab + Oxaliplatin
  Interventions: Drug: Irinotecan; Drug: Bevacizumab; Drug: Oxaliplatin
- Group 3 (Experimental): Group 3 = Irinotecan, Bevacizumab + Cetuximab
  Interventions: Drug: Irinotecan; Drug: Bevacizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Irinotecan — Starting dose of 35 mg/m^2 given through the catheter into your liver artery (hepatic artery infusion - HAI), continuously for 72 hours (Days 1 through 2 of each cycle).
  Other Names: CPT-11; Camptosar
Drug: Bevacizumab — 10 mg/Kg by vein on Days 1 and 15 of every 28 day cycle, over 90 minutes first cycle and over 30-60 minutes subsequent cycles.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Oxaliplatin — Starting dose 60 mg/m^2 by vein over 2 hours on Days 1 and 15 of every cycle.
  Other Names: Eloxatin
  Arms: Group 2
Drug: Cetuximab — 500 mg/m^2 by vein on Days 1 and 15 of every cycle. The first time given over 2 hours, all other cycles over 1 hour.
  Other Names: C225; Erbitux; IMC-C225
  Arms: Group 3

SUMMARY:
The goal of this clinical research study is to learn the highest tolerable dose of irinotecan that can be given directly into the liver, in combination with other drugs given by vein.

The other drug combinations given by vein include bevacizumab alone, bevacizumab plus oxaliplatin, and bevacizumab plus cetuximab.

This will be tested in patients with advanced solid tumors that have spread to the liver. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Irinotecan is designed to stop cancer cells from making new DNA (the genetic material of cells). This may cause cancer cells to die.

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels that supply nutrients necessary for tumor growth.

Oxaliplatin is designed to block new cancer cells from growing.

Cetuximab is designed to prevent or slow down the growth of cancer cells by blocking proteins inside cancer cells.

Study Arms and Dose Levels:

If you are found to be eligible to take part in this study, your doctor will assign you to a study arm. Your study arm will depend on the type of cancer, your Kirsten rat sarcoma (KRAS) test result (if applicable), and the drugs you have taken in the past.

* If you are in Arm A, you will receive irinotecan and bevacizumab.
* If you are in Arm B, you will receive irinotecan, bevacizumab, and oxaliplatin.
* If you are in Arm C, you will receive irinotecan, bevacizumab, and cetuximab.

The dose that you receive will depend on when you are enrolled in this study and the safety data that is available at that time. The first set of 3-6 participants to join each study arm will receive the lowest dose of the drug combination. The next set of 3-6 participants will receive a higher dose of the drug combination. Each new set of participants will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the drug combinations is found.

Once the highest tolerable dose is found for each arm, 14 participants with the tumor type that has responded well to a particular study drug combination will receive the study drugs at that dose level. These participants will be in the "expansion" arms.

Catheter Placement:

You will be hospitalized to receive the study drug combination. The morning after you enter the hospital, you will have a catheter placed in your right groin area. A catheter is a sterile flexible tube. It will be placed into a large artery (the blood vessel that carries blood to your liver) while the area is numbed with local anesthetic. Your doctor will explain this procedure to you in more detail, and you will be asked to sign a separate consent form for it.

After you return to your room, you will receive irinotecan as described below.

Study "cycles" will be repeated every 28 days. The catheter will be placed and removed during each cycle. Each time, you will lie in bed for the entire time that the catheter is in place. While the catheter is being removed, the study staff will apply pressure to your groin area for 15 minutes to stop the bleeding.

Study Drug Administration:

Irinotecan will be given through the catheter into your liver artery, continuously for 48hours (Days 1 through 2 of each cycle). Before every irinotecan dose, you will also receive drugs by vein to lower the risk of nausea, if your doctor thinks this is needed for routine care.

Bevacizumab will be given by vein once every 2 weeks. The first time you receive bevacizumab, it will be given over 90 minutes. If you tolerate it well, all other bevacizumab doses will be given over 30-60 minutes.

Oxaliplatin, if you receive it, will be given by vein over 2 hours once every 2 weeks. Before every oxaliplatin dose, you will also receive drugs by vein to lower the risk of nausea, if your doctor thinks this is needed for routine care.

Cetuximab, if you receive it, will be given by vein once every 2 weeks. The first time you receive cetuximab, it will be given over 2 hours. All other cetuximab doses will be given over 1 hour.

If you do not tolerate the study drug combination well, the doses that you receive may be lowered. If you experience certain side effects, your study drug doses may be delayed and the study cycle may be longer than 28 days.

You will be given standard drugs (heparin and diphenhydramine) to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

You will be in the hospital for about 5-7 days at the beginning of every cycle, until you recover from side effects that may occur. You will be seen by a doctor or "advanced practice" nurse every day while you are in the hospital.

At the beginning of each cycle and then once a week during each cycle, blood (about 1 tablespoon) will be drawn for routine tests. At the beginning of each cycle and then once every 4 weeks (or earlier if needed), you will have a physical exam.

You will have scans such as a chest x-ray, CT, MRI, and/or PET scan after every 2 cycles (8 weeks) or earlier if the study doctor thinks it is in your best interest, or the cancer gets worse. These scans are to check the status of the disease. If the study doctor thinks it is more appropriate for you, other types of scans may need to be performed. The study doctor will discuss these scans with you, and you may be asked to sign a separate consent form.

Additional Tests/Procedures for Some Participants:

If you experience severe diarrhea and/or low white blood cell counts while on this study, blood (about 2 teaspoons) will be drawn to test your DNA to find out if you may be at a higher risk of side effects from irinotecan. If the test shows that you may have a higher risk, then you will receive irinotecan at a lower dose level.

If you are in Arm C (which as discussed above, does not include colorectal cancer patients with a KRAS mutation), a leftover sample of tumor tissue will be tested for the KRAS mutation. If no leftover tumor tissue from an earlier procedure is available, and if your KRAS status is unknown, you will have a needle biopsy of a tumor performed. The tissue will be tested for the KRAS mutation. This procedure will be done on an appropriate tumor area that is able to be biopsied, and it may or may not be the liver tumor. This will be the doctor's decision.

Length of Study:

You may stay on study for as long as the disease has not gotten worse, the cancer has not gone away completely, and you have not experienced intolerable side effects. In any of those cases, you would be taken off study.

End-of-Study Visit:

About 28 days after your last dose of study drugs, you will have an end-of-study visit. At this visit, the following tests and procedures may be performed:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have an x-ray, CT scan, PET scan, or -MRI scan to check the status of the disease.

This is an investigational study. It is investigational to give irinotecan into a liver artery. The study drug combinations and dose levels are also investigational.

The study drugs are commercially available and FDA approved to treat the following:

* Irinotecan by vein -- colorectal cancer that is metastatic (has spread).
* Bevacizumab -- metastatic colorectal cancer, breast cancer, non small-cell lung cancer, and a type of brain cancer called glioblastoma multiforme.
* Cetuximab -- colorectal cancer, and head and neck cancer.
* Oxaliplatin -- colorectal cancer.

Up to 140 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed metastatic advanced cancers with liver involvement.
2. Patients should be refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that improves survival by at least three months, unless the drugs included in the regimen are part of their standard treatment.
3. Irinotecan will be dosed regardless of creatinine clearance. For oxaliplatin, serum creatinine </= 2.5 times the upper limit of normal or creatinine clearance >/= 40 is required.
4. Hepatic function: T. Bilirubin </= 3 mg/dl, ALT </= 5X upper limit of normal (ULN).
5. Adequate bone marrow function (ANC >/=1000 cells/uL; PLT >/= 100,000 cells/uL).
6. Patients must have been off previous chemotherapy or radiotherapy for the three weeks prior to entering this study. Six weeks will be required if the patient has received therapy which is known to have delayed toxicity (mitomycin or a nitrosurea). Five half-lives will be required for biologic/targeted therapies with short (<24 hour) half-lives and pharmacodynamic effects. Patients may have received palliative radiation immediately before (or during) treatment provided radiation is not to the only target lesion available.
7. All females in childbearing age MUST have a negative serum or urine pregnancy test unless prior hysterectomy or menopause (defined as age above 55 and six months without menstrual activity). Patients should not become pregnant or breast feed while on this study. Sexually active patients should use effective birth control.
8. Eastern Cooperative Oncology Group (ECOG) Performance status </= 2.

Exclusion Criteria:

1. Pregnant females.
2. Patients with colorectal cancer and K-RAS mutation will be excluded from the cetuximab arm.
3. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days.
4. Invasive procedures defined as follows: a. Major surgical procedure within 28 days prior to Day 1 therapy. b. Anticipation of need for major surgical procedures during the course of the study.
5. Patients receiving any other investigational agents.
6. Patients with bleeding diathesis (clinical bleeding, prothrombin time >/= 1.5 X upper institutional normal value, international normalized ratio (INR) >/=1.5, activated partial thromboplastin time aPTT >/= 1.5 X upper institutional normal value, NOT due to anticoagulation therapy), active gastric or duodenal ulcer.
7. Patients with history of bleeding CNS metastasis will be excluded from the trial.
8. Hypersensitivity to any of the drugs in a particular treatment arm.
9. Inability to complete informed consent process and adhere to protocol treatment plan and follow up requirements.
10. History of heparin-induced thrombocytopenia.
11. Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg on medication).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Doses (MTDs) | Evaulated with each 28 day cycle
  MTD is defined as the highest dose level at which ≥ 33% of patients have a DLT if >3 patients are treated at that dose level or > 33% have a DLT if ≤3 patients have been treated.
Dose-limiting toxicities (DLTs) | Evaulated with each 28 day cycle
  DLT defined as any grade 3 or 4 non-hematologic toxicity defined in NCI CTC v3.0, even if expected and believed related to study medications (except nausea and vomiting responsive to appropriate regimens or alopecia), any grade 4 hematologic toxicity lasting 2 weeks or longer (as defined by the NCI-CTCAE), despite supportive care; any grade 4 nausea or vomiting > 5 days despite maximum anti-nausea regimens, and any other grade 3 non-hematologic toxicity including symptoms/signs of vascular leak or cytokine release syndrome; or any severe or life-threatening complication or abnormality not defined in the NCI-CTCAE that is attributable to the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org